CLINICAL TRIAL: NCT02303574
Title: A PHASE I, RANDOMISED, SINGLE-BLIND, PLACEBO-CONTROLLED, 2-PART STUDY TO ASSESS THE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS AND FOOD EFFECT OF SINGLE AND MULTIPLE ORAL DOSES OF AZD7986 IN HEALTHY VOLUNTEERS.
Brief Title: Single + Multiple Ascending Dose and Food Effect Study of AZD7986 in Healthy Volunteers, PK, PD and Safety Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D6190C00001; 2014-004043-13 (EudraCT Number)
Record Dates: First submitted 2014-11-03; First posted 2014-12-01 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Safety, Pharmacokinetics, Pharmacodynamics, Food Effect
Keywords: AZD7986, Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Food Effect, First-in-human, Single Ascending Dose, Multiple Ascending Dose, Healthy Subjects
MeSH Terms: interventions — brensocatib; Solutions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD7986, single and mulltiple doses (Experimental): In Part 1 up to 8 cohorts with single doses starting with 5 mg AZD7986 as oral solution. In Part 2 up to 5 cohorts with multiple doses of AZD7986 as oral solution
  Interventions: Drug: AZD7986, oral solution, 1 to 50 mg/mL
- Placebo, single and multiple doses (Placebo Comparator): In Part 1 up to 8 cohorts and in Part 2 up to 5 cohorts with matching placebo to AZD7986 as oral solution
  Interventions: Drug: Placebo, oral solution

INTERVENTIONS:
Drug: AZD7986, oral solution, 1 to 50 mg/mL — Starting dose in single ascending dose part: 5 mg
  Arms: AZD7986, single and mulltiple doses
Drug: Placebo, oral solution — Matching placebo
  Arms: Placebo, single and multiple doses

SUMMARY:
This is a phase I, randomised, single-blind placebo-controlled, 2-part study to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and food effect of single and multiple oral doses of AZD7986 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent prior to any study specific procedures.
2. Healthy male or female subjects aged 18 to 50 years (inclusive) at screening with suitable veins for cannulation or repeated venepuncture.
3. Females must be of non-child-bearing potential, confirmed at screening by fulfilling one of the following criteria:

   * Post-menopausal defined as amenorrhoea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle stimulating hormone (FSH) and luteinising hormone (LH) levels in the post menopausal range.
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
4. Male subjects must be non fertile, i.e., surgically sterilised with documentation of azoospermia or must practice an effective contraceptive method to prevent pregnancies. Effective contraceptive methods are:

   * Sexual abstinence from before the first administration of the IMP until 3 months after final administration of the IMP, only if this is in line with the preferred and usual lifestyle of the subject.
   * Use of a condom plus spermicide agent in addition to having their partner use another acceptable method (oral or injectable hormonal contraceptives, contraceptive patch, intrauterine devices, vaginal hormonal rings, vaginal diaphragm or cervical caps) from before the first administration of the IMP until 3 months after final administration of the IMP.
   * Subject's sexual partner is of non childbearing potential, i.e., post menopausal or surgically sterilised (e.g., tubal ligation, hysterectomy in medical history).
5. Have a body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive at screening.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
* Subject has increased risk of infection:

  * History and/or presence of tuberculosis (TB); positive result for interferon gamma release assay (IGRA) (i.e., QuantiFERON TB-Gold), subjects who have resided in regions where tuberculosis and mycosis are endemic during 90 days before screening, or who intend to visit such a region during the duration of the study i.e. deserts areas, Eastern Europe, Central and South America, Africa except Egypt, Russia, Asia, Indonesia
  * Oral body temperature of > 37.7°C on Day -1, or as judged by the Investigator.
  * Blood neutrophil count < 1.7 x109/L (Screening and Day -1 morning sample).
  * Is in high risk-group for HIV infection within the last 6 months (i.e., men who have had unprotected sex with men, women who have had sex without a condom with men who have sex with men, people who have had sex without a condom with a person who has lived or travelled in Africa, people who inject drugs, people who have had sex without a condom with somebody who has injected drugs, people who have caught another sexually transmitted infection, people who have received a blood transfusion while in Africa, eastern Europe, the countries of the former Soviet Union, Asia or central and southern America).
  * Other latent or chronic infections (e.g., recurrent sinusitis, genital or ocular herpes, urinary tract infection) or at risk of infection (surgery, trauma, or significant infection) within 90 days of screening, or history of skin abscesses within 90 days of screening.
  * Clinically significant lower respiratory tract infection not resolved within 4 weeks prior to screening, as determined by the Investigator.
  * Volunteers with active malignancy or neoplastic disease in the previous 5 years other than superficial basal cell carcinoma.
  * Disease history suggesting abnormal immune function.
  * Volunteers who have received live or live-attenuated vaccine in the 4 weeks prior to dosing.
  * High-sensitivity C-reactive protein above upper limit of laboratory reference range at screening and on Day -1.
* Some subjects lacking functional dipeptidyl peptidase 1 (DPP1) enzyme have been described to have periodontitis and palmoplantar hyperkeratosis:

  * For Part 1a and Part 1b: Subjects with signs of current gingivitis/periodontitis. Gingival evaluation (by inspection) will be performed by a dental hygienist or trained study physician.
  * For Part 2: Subjects with a history of recurring gingivitis/periodontitis or signs of current gingivitis/periodontitis. Gingival evaluation will be performed by a dental hygienist or trained study physician. Evaluation of bleeding propensity due to gingivitis will be performed by using dental hygienist instrumentation. Exact measurement of gum pockets is not needed.
  * Subjects with a history of hyperkeratosis or erythema in palms or soles.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2016-08-03 (Actual); Study Completion 2016-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, Dr, Principal Investigator — PAREXEL Early Phase Clinical Unit, Level 7, Northwick Park Hospital, Watford Road, Harrow, Middlesex, HA1 3UJ, United Kingdom; Bengt Larsson, Study Chair — AstraZeneca
Locations (1):
- Research Site, Harrow, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at PAREXEL Early Phase Clinical Unit London, Level 7, Northwick Park Hospital in London. Healthy male and female participants were enrolled.
Pre-assignment Details: In Part 1 and Part 2, participants underwent a screening visit within 28 days before receiving the first dose of investigational medicinal product (IMP). Participants were admitted to the study centre 1 day before administration of the IMP (Day -1).
Groups:
- AZD7986 5 mg (Fasted State) - SAD: Participants received single dose of oral solution of AZD7986 5mg on Day 1 in fasted state.
- AZD7986 15 mg (Fasted State) - SAD: Participants received single dose of oral solution of AZD7986 15mg on Day 1in fasted state.
- AZD7986 35 mg (Fasted State) - SAD: Participants received single dose of oral solution of AZD7986 35mg on Day 1 in fasted state.
- AZD7986 50 mg (Fasted State) - SAD: Participants received single dose of oral solution of AZD7986 50mg on Day 1 in fasted state.
- AZD7986 65 mg (Fasted State) - SAD: Participants received single dose of oral solution of AZD7986 65mg on Day 1 in fasted state.
- AZD7986 35 mg (Fed State) - SAD: Participants of Cohorts 3 from Part 1a received single dose of oral solution of AZD7986 35 mg on Day 1 in fed state after a washout of at least 7 days.
- AZD7986 10 mg - MAD: Participants received single dose (morning) of oral solution of AZD7986 10 mg for 28 days (fasted or fed state, depending on Part 1b results). Participants were fasted until 1 hour after dosing when a light breakfast was provided.
- AZD7986 25 mg - MAD: Participants received single dose (morning) of oral solution of AZD7986 25 mg for 28 days (fasted or fed state, depending on Part 1b results). Participants were fasted until 1 hour after dosing when a light breakfast was provided.
- AZD7986 40 mg - MAD: Participants received single dose (morning) of oral solution of AZD7986 40 mg for 28 days (fasted or fed state, depending on Part 1b results). Participants were fasted until 1 hour after dosing when a light breakfast was provided.
- Placebo: Randomized participants received orally AZD7986 matching placebo oral solution.
Period: Part 1a (Fasted State)- SAD
Arm/Group | AZD7986 5 mg (Fasted State) - SAD | AZD7986 15 mg (Fasted State) - SAD | AZD7986 35 mg (Fasted State) - SAD | AZD7986 50 mg (Fasted State) - SAD | AZD7986 65 mg (Fasted State) - SAD | AZD7986 35 mg (Fed State) - SAD | AZD7986 10 mg - MAD | AZD7986 25 mg - MAD | AZD7986 40 mg - MAD | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 15 (Participants received AZD7986 matching placebo on Day 1 in fasted state.)
Completed | 6 | 6 | 5 | 6 | 6 | 0 | 0 | 0 | 0 | 15
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1b (Fed State) - SAD
Arm/Group | AZD7986 5 mg (Fasted State) - SAD | AZD7986 15 mg (Fasted State) - SAD | AZD7986 35 mg (Fasted State) - SAD | AZD7986 50 mg (Fasted State) - SAD | AZD7986 65 mg (Fasted State) - SAD | AZD7986 35 mg (Fed State) - SAD | AZD7986 10 mg - MAD | AZD7986 25 mg - MAD | AZD7986 40 mg - MAD | Placebo
Started | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 3 (Participants received AZD7986 matching placebo on Day 1 in fed state.)
Completed | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 - Multiple Ascending Dose (MAD)
Arm/Group | AZD7986 5 mg (Fasted State) - SAD | AZD7986 15 mg (Fasted State) - SAD | AZD7986 35 mg (Fasted State) - SAD | AZD7986 50 mg (Fasted State) - SAD | AZD7986 65 mg (Fasted State) - SAD | AZD7986 35 mg (Fed State) - SAD | AZD7986 10 mg - MAD | AZD7986 25 mg - MAD | AZD7986 40 mg - MAD | Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 10 | 12 (Participants took AZD7986 matching placebo for 28 days (fasted/fed state, based on part 1b results))
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 7 | 10 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo - Part 1a (Fasted): Randomized participants received orally AZD7986 matching placebo oral solution on Day 1 in fasted state.
- Placebo - Part 1b (Fed State): Randomized participants received orally AZD7986 matching placebo oral solution on Day 1 in fed state.
- Placebo - Part 2: Randomized participants received orally AZD7986 matching placebo oral solution for 28 days (fasted/fed state, based on part 1b results).
- Total: Total of all reporting groups
Arm/Group | AZD7986 5 mg (Fasted State) - SAD | AZD7986 15 mg (Fasted State) - SAD | AZD7986 35 mg (Fasted State) - SAD | AZD7986 50 mg (Fasted State) - SAD | AZD7986 65 mg (Fasted State) - SAD | AZD7986 35 mg (Fed State) - SAD | AZD7986 10 mg - MAD | AZD7986 25 mg - MAD | AZD7986 40 mg - MAD | Placebo - Part 1a (Fasted) | Placebo - Part 1b (Fed State) | Placebo - Part 2 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 8 | 10 | 15 | 3 | 12 | 89
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All randomized participants who received at least one dose of IMP were included for the presentation of all demographic data.
  Years
    Part 1a: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30
    Part 1a | 28.5 (5.39) | 29.7 (8.78) | 26.2 (3.66) | 32.2 (10.5) | 29.7 (6.65) |  |  |  |  |  |  |  | 29.2 (7.14)
    Part 1b: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 5
    Part 1b |  |  |  |  |  | 26.6 (3.91) |  |  |  |  |  |  | 26.6 (3.91)
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 10 | 0 | 0 | 0 | 24
    Part 2 |  |  |  |  |  |  | 30.7 (5.65) | 38.4 (7.25) | 34.4 (9.17) |  |  |  | 34.8 (8.05)
    Part 1a Placebo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 15
    Part 1a Placebo |  |  |  |  |  |  |  |  |  | 29.9 (7.24) |  |  | 29.9 (7.24)
    Part 1b Placebo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3
    Part 1b Placebo |  |  |  |  |  |  |  |  |  |  | 28.7 (8.5) |  | 28.7 (8.5)
    Part 2 Placebo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12
    Part 2 Placebo |  |  |  |  |  |  |  |  |  |  |  | 36.2 (7.2) | 36.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All randomised subjects who received at least one dose of IMP were included for the presentation of all demographic data.
  Participants
    Part 1a: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 45
    Part 1a: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part 1a: Male | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 45
    Part 1b: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 3 | 0 | 8
    Part 1b: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part 1b: Male | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 3 | 0 | 8
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 10 | 0 | 0 | 12 | 36
    Part 2: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part 2: Male | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 8 | 10 | 0 | 0 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of AZD7986 by Assessment of the Number of Adverse Events (AEs) Following Administration of Oral Solution in Single Ascending Dose (SAD - Part 1a and 1b) and Multiple Ascending Doses (MAD -Part 2)
Description: To investigate the safety and tolerability of AZD7986 by assessment of AEs (non-serious and serious) following administration of oral solution in SAD (Part 1a - fasted state and 1b - fed state) and MAD (Part 2)
Time Frame: Part 1a and 1b: Day -1, Day 1 to Day 3 (spontaneous, at pre-dose, 3, 12, 24, 48 and 72 hours [h] post-dose), Day 4, Day 5 and follow-up (7-10 days after dosing [not for participants included in Part 1b]); Part 2: Day -1, Day 1 to Day 21/28 and follow-up
Population: All randomized subjects who received at least one dose of IMP were included in the safety analysis for the study.
Measure: Number; unit: Participants
Groups:
- Part 1a (Fasted State) - Single Ascending Dose (SAD): Participants received single dose of oral solution of AZD7986 at 5 ascending doses (5mg, 15mg, 35mg, 50mg and 65mg) on Day 1 in fasted state with 6 participants in each dose level.
- Part 1b (Fed State) - SAD: 5 Participants of Cohort 3 from Part 1a received single dose of oral solution of AZD7986 35mg on Day 1 in fed state after a washout of at least 7 days.
- Part 2 - Multiple Ascending Dose (MAD): 24 participants (6 in Cohort 1-10mg, 8 in Cohort 2- 25mg and 10 in Cohort 3-40mg) received once daily dose of oral solution of AZD7986 in the morning for 28 days. Participants were fasted until 1 hour after dosing when a light breakfast was provided.
- Placebo - Part 1a (Fasted State)- SAD: 3 participants per dose level received single dose of oral solution of placebo in Part 1a in fasted state on Day 1
- Placebo - Part 1b (Fed State) - SAD: 3 participants of Cohort 3 from Part 1a received single dose of oral solution of placebo 35mg on Day 1 in fed state after a washout of at least 7 days.
- Placebo - Part 2 - MAD: 12 participants (randomized 6:3, 8:3 and 10:4/10:6/12:4) received once daily dose of oral solution of Placebo in the morning for 28 days. Participants were fasted until 1 hour after dosing when a light breakfast was provided.
Arm/Group | Part 1a (Fasted State) - Single Ascending Dose (SAD) | Part 1b (Fed State) - SAD | Part 2 - Multiple Ascending Dose (MAD) | Placebo - Part 1a (Fasted State)- SAD | Placebo - Part 1b (Fed State) - SAD | Placebo - Part 2 - MAD
Number analyzed (Participants) | 30 | 5 | 24 | 15 | 3 | 12
Participants
  Any AE | 8 | 2 | 23 | 8 | 1 | 8
  Any AE with outcome = death | 0 | 0 | 0 | 0 | 0 | 0
  Any serious adverse event (SAE) (including death) | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of AZD7986 | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Rate and Extent of Absorption AZD7986 by Assessment of the Area Under the Plasma Concentration Versus Time Curve, From Time Zero to the Time of the Last Quantifiable Concentration (AUC(0-last)) for Part 1a and 1b - SAD
Description: To assess the area under the plasma concentration versus time curve, from time zero to the time of the last quantifiable analyte concentration (AUC(0-last)) for Part 1a (fasted state) and 1b (fed state) - SAD
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 h); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: The pharmacokinetic analysis (PK) analysis set consisted of all subjects in the safety analysis set who received at least 1 dose of AZD7986 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h·nmol/L
Groups:
- AZD7986 5mg - Part 1a (Fasted State) - SAD: Participants received single dose of oral solution of AZD7986 5mg on Day 1 in fasted state.
- AZD7986 15mg - Part 1a (Fasted State) - SAD: Participants received single dose of oral solution of AZD7986 15mg on Day 1.
- AZD7986 35mg - Part 1a (Fasted State) - SAD: Participants received single dose of oral solution of AZD7986 35mg on Day 1 in fasted state.
- AZD7986 50mg - Part 1a (Fasted State) - SAD: Participants received single dose of oral solution of AZD7986 50mg on Day 1
- AZD7986 65mg - Part 1a (Fasted State) - SAD: Participants received single dose of oral solution of AZD7986 65mg on Day 1
- AZD7986 35mg - Part 1b (Fed State) - SAD: Participants received single dose of oral solution of AZD7986 35mg on Day 1.
Arm/Group | AZD7986 5mg - Part 1a (Fasted State) - SAD | AZD7986 15mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 50mg - Part 1a (Fasted State) - SAD | AZD7986 65mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
h·nmol/L | 839.0 (48.3) | 3855 (9.3) | 12430 (18.3) | 16470 (22.7) | 22880 (21.2) | 10790 (20.2)

3. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of the Area Under the Plasma Concentration Versus Time Curve, From Time Zero to the Time of the Last Quantifiable Analyte Concentration (AUC(0-last)) for Part 2 - MAD
Description: To assess the area under the plasma concentration versus time curve, from time zero to the time of the last quantifiable analyte concentration (AUC(0-last)) following a single AZD7986 dose on Day 1 and daily dosing on Days 21 or 28 at 10, 25 and 40 mg in Part 2
Time Frame: Day 1 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 8, 9, 12, 24 h); Day 21 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 8, 9, 12, 24, 72, 96 h) and Day 28
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h·nmol/L
Groups:
- AZD7986 10mg - Day 1 - Part 2 - MAD; AZD7986 10mg - Day 21 - Part 2 - MAD: Participants received single dose of oral solution of AZD7986 10mg on Day 1 and daily dosing on Days 21 or 28 in fasted state.
- AZD7986 25mg - Day 1 - Part 2 - MAD; AZD7986 25mg - Day 28 - Part 2 - MAD: Participants received single dose of oral solution of AZD7986 25mg on Day 1 and daily dosing on Days 21 or 28 in fasted state.
- AZD7986 40mg - Day 1 - Part 2 - MAD; AZD7986 40mg - Day 28 - Part 2 - MAD: Participants received single dose of oral solution of AZD7986 40mg on Day 1 and daily dosing on Days 21 or 28 I fasted state.
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
h·nmol/L | 1278 (18.9) [0.50 to 1.00] | 3256 (15.9) [0.53 to 2.00] | 6427 (31.0) [0.53 to 1.50] | 5135 (49.4) | 14320 (39.5) | 29550 (53.5)

4. Primary Outcome: Rate and Extent of Absorption AZD7986 by Assessment of the Area Under Plasma Concentration-time Curve From Zero Extrapolated to Infinity (AUC) for Part 1a and 1b - SAD
Description: To assess the area under plasma concentration-time curve from zero extrapolated to infinity (AUC) for Part 1a (fasted state) and 1b (fed state) - SAD. AUC was estimated by AUC(0 last) + Clast/λz where Clast was the last observed quantifiable concentration.
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 h); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h·nmol/L
Arm/Group | AZD7986 5mg - Part 1a (Fasted State) - SAD | AZD7986 15mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 50mg - Part 1a (Fasted State) - SAD | AZD7986 65mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
h·nmol/L | 915.3 (46.1) | 4165 (10.8) | 13230 (19.6) | 17590 (25.2) | 24710 (21.5) | 11550 (22.6)
Statistical Analysis 1: Comparison: AZD7986 5mg - Part 1a (Fasted State) - SAD vs AZD7986 15mg - Part 1a (Fasted State) - SAD vs AZD7986 35mg - Part 1a (Fasted State) - SAD vs AZD7986 50mg - Part 1a (Fasted State) - SAD vs AZD7986 65mg - Part 1a (Fasted State) - SAD; Test type: Other — Dose proportionality was analyzed by power model. Slope parameter was obtained via linear least squares; Slope = 1.287, 95% CI 2-sided [1.183 to 1.391], Standard Error of Mean 0.05085
Statistical Analysis 2: Comparison: AZD7986 35mg - Part 1a (Fasted State) - SAD vs AZD7986 35mg - Part 1b (Fed State) - SAD; Test type: Other — Effect of food analysis by linear mixed effects ANOVA model with fixed effect of fasting status; Ratio (%) = 90.72, 90% CI 2-sided [83.72 to 98.31]

5. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of the Area Under Plasma Concentration-time Curve From Zero Extrapolated to Infinity (AUC) for Part 2 - MAD
Description: To assess the area under plasma concentration-time curve from zero extrapolated to infinity (AUC) following a single AZD7986 dose on Day 1 and daily dosing on Days 21 or 28 at 10, 25 and 40 mg in Part 2. Note: Day 1 data calculated over a 24 hour period and was therefore not comparable with the Day 21 and Day 28 data
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h·nmol/L
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
h·nmol/L | 1778 (21.3) [0.50 to 1.00] | 4957 (19.5) [0.53 to 2.00] | 9866 (35.8) [0.53 to 1.50] | 5565 (54.3) | 16660 (44.2) | 33220 (58.5)
Statistical Analysis 1: Comparison: AZD7986 10mg - Day 1 - Part 2 - MAD vs AZD7986 10mg - Day 21 - Part 2 - MAD; Test type: Other — Time dependency was assessed via linear mixed effects ANOVA model with fixed effects of dose level, day and dose-level-by-day interaction; Ratio (%) = 159.40, 90% CI 2-sided [140.61 to 180.70]
Statistical Analysis 2: Comparison: AZD7986 25mg - Day 1 - Part 2 - MAD vs AZD7986 25mg - Day 28 - Part 2 - MAD; Test type: Other — [test comment as in outcome 5, analysis 1]; Ratio (%) = 151.82, 90% CI 2-sided [138.23 to 166.74]
Statistical Analysis 3: Comparison: AZD7986 40mg - Day 1 - Part 2 - MAD vs AZD7986 40mg - Day 28 - Part 2 - MAD; Test type: Other — [test comment as in outcome 5, analysis 1]; Ratio (%) = 158.68, 90% CI 2-sided [146.67 to 171.67]

6. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval (AUCτ) for Part 2 - MAD
Description: To assess area under the plasma concentration-time curve from time zero to the end of the dosing interval (AUCτ) following a single AZD7986 dose on Day 1 and daily dosing on Days 21 or 28 at 10, 25 and 40 mg in Part 2. AUCτ: AUC from time zero to 24 hours post-dose presented on Day1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h·nmol/L
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
h·nmol/L | 1277 (18.9) [0.50 to 1.00] | 3259 (15.9) [0.53 to 2.00] | 6433 (31.0) [0.53 to 1.50] | 2834 (35.1) | 7499 (27.4) | 15660 (43.3)
Statistical Analysis 1: Comparison: AZD7986 10mg - Day 1 - Part 2 - MAD vs AZD7986 25mg - Day 1 - Part 2 - MAD vs AZD7986 40mg - Day 1 - Part 2 - MAD vs AZD7986 10mg - Day 21 - Part 2 - MAD vs AZD7986 25mg - Day 28 - Part 2 - MAD vs AZD7986 40mg - Day 28 - Part 2 - MAD; Test type: Other — Dose proportionality was analyzed by power model. Slope parameter was obtained via linear least squares; Slope = 1.228, 95% CI 2-sided [0.9513 to 1.504], Standard Error of Mean 0.1329
Statistical Analysis 2: Comparison: AZD7986 10mg - Day 1 - Part 2 - MAD vs AZD7986 10mg - Day 21 - Part 2 - MAD; Test type: Other — ime dependency was assessed via linear mixed effects ANOVA model with fixed effects of dose level, day and dose-level-by-day interaction; Ratio (%) = 159.40, 90% CI 2-sided [140.61 to 180.70]
Statistical Analysis 3: Comparison: AZD7986 25mg - Day 1 - Part 2 - MAD vs AZD7986 25mg - Day 28 - Part 2 - MAD; Test type: Other — [test comment as in outcome 6, analysis 2]; Ratio (%) = 151.82, 90% CI 2-sided [138.23 to 166.74]
Statistical Analysis 4: Comparison: AZD7986 40mg - Day 1 - Part 2 - MAD vs AZD7986 40mg - Day 28 - Part 2 - MAD; Test type: Other — [test comment as in outcome 6, analysis 2]; Ratio (%) = 158.68, 90% CI 2-sided [146.67 to 171.67]

7. Primary Outcome: Rate and Extent of Absorption AZD7986 by Assessment of the Observed Maximum Plasma Concentration (Cmax) for Part 1a and 1b - SAD
Description: To assess the observed maximum plasma concentration (Cmax) for Part 1a (fasted state) and 1b (fed state) - SAD. Cmax was taken directly from the individual concentration-time curve
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 h); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD7986 5mg - Part 1a (Fasted State) - SAD | AZD7986 15mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 50mg - Part 1a (Fasted State) - SAD | AZD7986 65mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
nmol/L | 50.74 (47.2) | 202.3 (16.0) | 668.1 (26.7) | 1035 (11.5) | 1358 (24.2) | 434.8 (14.0)
Statistical Analysis 1: Comparison: AZD7986 5mg - Part 1a (Fasted State) - SAD vs AZD7986 15mg - Part 1a (Fasted State) - SAD vs AZD7986 35mg - Part 1a (Fasted State) - SAD vs AZD7986 50mg - Part 1a (Fasted State) - SAD vs AZD7986 65mg - Part 1a (Fasted State) - SAD; Dose proportionality was analyzed by power model. Slope parameter was obtained via linear least squares; Test type: Other; Slope = 1.302, 95% CI 2-sided [1.198 to 1.406], Standard Error of Mean 0.05056
Statistical Analysis 2: Comparison: AZD7986 35mg - Part 1a (Fasted State) - SAD vs AZD7986 35mg - Part 1b (Fed State) - SAD; Test type: Other — Effect of food analysis by linear mixed effects ANOVA model with fixed effect of fasting status; Ratio (%) = 64.14, 90% CI 2-sided [55.07 to 74.70]

8. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of the Observed Maximum Plasma Concentration (Cmax) for Part 2 - MAD
Description: To assessthe observed maximum plasma concentration (Cmax) following a single AZD7986 dose on Day 1 and daily dosing on Days 21 or 28 at 10, 25 and 40 mg in Part 2. Cmax was taken directly from the individual concentration-time curve
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
nmol/L | 138.6 (18.3) [0.50 to 1.00] | 350.9 (19.3) [0.53 to 2.00] | 672.0 (37.0) [0.53 to 1.50] | 246.3 (26.2) | 598.1 (15.5) | 1235 (37.7)
Statistical Analysis 1: Comparison: AZD7986 10mg - Day 1 - Part 2 - MAD vs AZD7986 25mg - Day 1 - Part 2 - MAD vs AZD7986 40mg - Day 1 - Part 2 - MAD vs AZD7986 10mg - Day 21 - Part 2 - MAD vs AZD7986 25mg - Day 28 - Part 2 - MAD vs AZD7986 40mg - Day 28 - Part 2 - MAD; Test type: Other — Dose proportionality was analyzed by power model. Slope parameter was obtained via linear least squares; Slope = 1.157, 95% CI 2-sided [0.9285 to 1.385], Standard Error of Mean 0.1098

9. Primary Outcome: Rate and Extent of Absorption AZD7986 by Assessment of the Time to Reach Maximum Observed Concentration (Tmax) for Part 1a and 1b - SAD
Description: To assess the time to reach maximum observed concentration (tmax) for Part 1a (fasted state) and 1b (fed state) - SAD; tmax was taken directly from the individual concentration-time curve
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 h); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour
Arm/Group | AZD7986 5mg - Part 1a (Fasted State) - SAD | AZD7986 15mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 50mg - Part 1a (Fasted State) - SAD | AZD7986 65mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
Hour | 0.50 (47.2) [0.50 to 1.00] | 0.75 (16.0) [0.53 to 2.00] | 0.75 (26.7) [0.53 to 1.50] | 0.64 (11.5) [0.52 to 0.75] | 0.75 (24.2) [0.52 to 1.98] | 4.00 (14.0) [3.00 to 4.98]

10. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of the Time to Reach Maximum Observed Concentration (Tmax) for Part 2 - MAD
Description: To assess the time to reach maximum observed concentration (tmax) following a single AZD7986 dose on Day 1 and daily dosing on Days 21 or 28 at 10, 25 and 40 mg in Part 2; tmax was taken directly from the individual concentration-time curve
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
Hour | 1.51 (21.3) [0.52 to 1.53] | 0.75 (19.5) [0.53 to 2.00] | 0.75 (35.8) [0.52 to 1.50] | 1.50 [0.75 to 1.50] | 0.75 [0.52 to 2.00] | 1.12 [0.53 to 1.50]

11. Primary Outcome: Rate and Extent of Absorption AZD7986 by Assessment of the Apparent Terminal Elimination Half-life (t½.λz) for Part 1a and 1b - SAD
Description: To assess the half life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½.λz) for Part 1a (fasted state) and 1b (fed state) - SAD
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 h); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | AZD7986 5mg - Part 1a (Fasted State) - SAD | AZD7986 15mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 50mg - Part 1a (Fasted State) - SAD | AZD7986 65mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
Hour | 19.96 (3.416) [0.50 to 1.00] | 25.92 (4.452) [0.53 to 2.00] | 23.80 (3.328) [0.53 to 1.50] | 24.52 (5.836) [0.52 to 0.75] | 25.50 (7.254) [0.52 to 1.98] | 24.24 (4.259) [3.00 to 4.98]

12. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of the Apparent Terminal Elimination Half-life (t½.λz) for Part 2 - MAD
Description: To assess the apparent terminal elimination half-life (t½.λz) following a single AZD7986 dose on Day 1 and daily dosing on Days 21 or 28 at 10, 25 and 40 mg in Part 2; tmax was taken directly from the individual concentration-time curve. Note: Day 1 data were calculated over a 24 hour period and was therefore not comparable with the Day 21 and Day 28 data
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
Hour | 12.82 (1.477) [0.52 to 1.53] | 14.85 (2.244) [0.53 to 2.00] | 15.85 (4.132) [0.52 to 1.50] | 25.85 (5.501) | 33.78 (10.31) | 30.04 (5.483)

13. Primary Outcome: Rate and Extent of Absorption AZD7986 by Assessment of the Mean Residence Time (MRT) for Part 1a and 1b - SAD
Description: To assess the mean residence time (MRT) for Part 1a (fasted state) and 1b (fed state) - SAD
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 h); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | AZD7986 5mg - Part 1a (Fasted State) - SAD | AZD7986 15mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 50mg - Part 1a (Fasted State) - SAD | AZD7986 65mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
Hour | 27.03 (4.373) [0.50 to 1.00] | 34.94 (5.863) [0.53 to 2.00] | 32.15 (5.003) [0.53 to 1.50] | 32.19 (8.360) [0.52 to 0.75] | 33.76 (10.35) [0.52 to 1.98] | 33.73 (6.429) [3.00 to 4.98]

14. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of Mean Residence Time (MRT) for Part 2 - MAD
Description: To assess the mean residence time (MRT) following a single AZD7986 dose on Day 1 and daily dosing on Days 21 or 28 at 10, 25 and 40 mg in Part 2
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
Hour | 18.56 (2.245) [0.52 to 1.53] | 21.84 (3.067) [0.53 to 2.00] | 22.64 (5.844) [0.52 to 1.50] | 33.73 (9.663) | 40.16 (10.58) | 37.46 (8.157)

15. Primary Outcome: Rate and Extent of Absorption AZD7986 by Assessment of the Apparent Clearance (CL/F) for Part 1a and 1b - SAD
Description: To assess the apparent clearance (CL/F) for Part 1a (fasted state) and 1b (fed state) - SAD; CL/F for parent drug was estimated as dose divided by AUC
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 h); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litre/Hour
Arm/Group | AZD7986 5mg - Part 1a (Fasted State) - SAD | AZD7986 15mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 50mg - Part 1a (Fasted State) - SAD | AZD7986 65mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
Litre/Hour | 14.23 (7.577) [0.50 to 1.00] | 8.606 (0.9321) [0.53 to 2.00] | 6.395 (1.281) [0.53 to 1.50] | 6.938 (1.777) [0.52 to 0.75] | 6.371 (1.317) [0.52 to 1.98] | 7.363 (1.810) [3.00 to 4.98]

16. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of the Apparent Clearance (CL/F) for Part 2 - MAD
Description: To assess the apparent clearance (CL/F) following a single AZD7986 dose on Day 1 and daily dosing on Days 21 or 28 at 10, 25 and 40 mg in Part 2; CL/F for parent drug was estimated as dose divided by AUC
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litre/Hour
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
Litre/Hour | 13.61 (2.665) [0.52 to 1.53] | 12.20 (2.485) [0.53 to 2.00] | 10.24 (4.206) [0.52 to 1.50] | 8.786 (2.772) | 8.165 (2.025) | 6.577 (2.867)

17. Primary Outcome: Rate and Extent of Absorption AZD7986 by Assessment of the Apparent Volume of Distribution (Vz/F) for Part 1a and 1b - SAD
Description: To assess the apparent volume of distribution (Vz/F) for Part 1a (fasted state) and 1b (fed state) - SAD; Vz/F at terminal phase (extravascular administration) was estimated by dividing the apparent clearance (CL/F) by λz
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 h); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | AZD7986 5mg - Part 1a (Fasted State) - SAD | AZD7986 15mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 50mg - Part 1a (Fasted State) - SAD | AZD7986 65mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
Litre | 385.1 (129.6) [0.50 to 1.00] | 318.8 (46.72) [0.53 to 2.00] | 215.8 (29.62) [0.53 to 1.50] | 236.8 (39.64) [0.52 to 0.75] | 231.0 (67.56) [0.52 to 1.98] | 249.5 (24.96) [3.00 to 4.98]

18. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of the Apparent Volume of Distribution (Vz/F) for Part 2 - MAD
Description: To assess the the apparent volume of distribution (Vz/F) following a single AZD7986 dose on Day 1 and daily dosing on Days 21 or 28 at 10, 25 and 40 mg in Part 2; Vz/F at terminal phase (extravascular administration) was estimated by dividing the apparent clearance (CL/F) by λz
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
Litre | 248.9 (38.94) [0.52 to 1.53] | 256.7 (36.11) [0.53 to 2.00] | 222.7 (65.93) [0.52 to 1.50] | 311.8 (56.96) | 393.2 (163.1) | 269.6 (79.13)

19. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of the Accumulation Ratio for (Rac(AUC(0-τ)) for Part 2 - MAD
Description: To assess the accumulation ratio for (Rac(AUC(0-τ)) following a single AZD7986 dose on Day 1 and daily dosing on Days 21 or 28 at 10, 25 and 40 mg in Part 2; estimated as AUC(0-τ) Day 21/AUC(0-24) Day 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
Ratio | NA (NA) — NA - Not applicable. Not assessed for Day 1 | NA (NA) — NA - Not applicable. Not assessed for Day 1 | NA (NA) — NA - Not applicable. Not assessed for Day 1 | 2.257 (0.4560) | 2.330 (0.4828) | 2.476 (0.4521)

20. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of the Accumulation Ratio for Cmax (Rac(Cmax)) for Part 2 - MAD
Description: To assess the accumulation ratio for Cmax (Rac(Cmax)) following a single AZD7986 dose on Day 1 and daily dosing on Days 21 or 28 at 10, 25 and 40 mg in Part 2; estimated as Cmax Day 21/Cmax Day 1
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
Ratio | NA (NA) — NA - Not applicable. Not assessed for Day 1 | NA (NA) — NA - Not applicable. Not assessed for Day 1 | NA (NA) — NA - Not applicable. Not assessed for Day 1 | 1.799 (0.3084) | 1.667 (0.2007) | 1.881 (0.4015)

21. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of the Temporal Change Parameter (TCP) for Part 2 - MAD
Description: To assess the temporal change parameter (TCP) following a single AZD7986 dose on Day 1 and daily dosing on Days 21 or 28 at 10, 25 and 40 mg in Part 2; estimated as AUC(0-τ) Day 21/AUC Day 1, if extrapolated part was less than 20%
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
Ratio | NA (NA) — NA - Not applicable. Not assessed for Day 1 | NA (NA) — NA - Not applicable. Not assessed for Day 1 | NA (NA) — NA - Not applicable. Not assessed for Day 1 | 1.610 (0.2539) | 1.535 (0.2479) | 1.599 (0.2082)

22. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of Urine PK Parameter (Cumulative Amount of Analyte Excreted From 0 to 48 Hours (CumAe0-48)) Following Administration of Single Dose Oral Solution for Part 1a and 1b - SAD
Description: To assess cumulative amount of analyte excreted from 0 to 48 hours (CumAe0-48) after single dose administration of AZD7986 oral solution in Part 1a (fasted state) and 1b (fed state)
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 h); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | AZD7986 5mg - Part 1a (Fasted State) - SAD | AZD7986 15mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 50mg - Part 1a (Fasted State) - SAD | AZD7986 65mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
nmol | 1318 (348.5) [0.50 to 1.00] | 4820 (1096) [0.53 to 2.00] | 16530 (2145) [0.53 to 1.50] | 19660 (4521) [0.52 to 0.75] | 27770 (10200) [0.52 to 1.98] | 18420 (2554) [3.00 to 4.98]

23. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of Urine PK Parameter (Percentage of Dose Excreted Unchanged Into the Urine From 0 to 48 Hours (Cumfe0-48)) Following Administration of Single Dose Oral Solution for Part 1a and 1b - SAD
Description: To assess percentage of dose excreted unchanged into the urine from 0 to 48 hours (Cumfe0-48) after single dose administration of AZD7986 oral solution in Part 1a (fasted state) and 1b (fed state)
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 h); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of dose excreted unchanged
Arm/Group | AZD7986 5mg - Part 1a (Fasted State) - SAD | AZD7986 15mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 50mg - Part 1a (Fasted State) - SAD | AZD7986 65mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
Percentage of dose excreted unchanged | 11.09 (2.931) | 13.51 (3.074) | 19.86 (2.578) | 16.53 (3.802) | 17.97 (6.598) | 22.13 (3.069)

24. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of Urine PK Parameter (Renal Clearance From 0 to 48 Hours (CLR0-48)) Following Administration of Single Dose Oral Solution for Part 1a and 1b - SAD
Description: To assess renal clearance from 0 to 48 hours (CLR0-48) after single dose administration of AZD7986 oral solution in Part 1a (fasted state) and 1b (fed state)
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 h); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | AZD7986 5mg - Part 1a (Fasted State) - SAD | AZD7986 15mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 50mg - Part 1a (Fasted State) - SAD | AZD7986 65mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5
Liter/hour | 1.734 (0.368) | 1.544 (0.2898) | 1.619 (0.2101) | 1.430 (0.1561) | 1.477 (0.5187) | 2.097 (0.1921)

25. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of Urine PK (Cumulative Amount of Analyte Excreted From 0 to 24 Hours (CumAe0-24)) Parameters for Part 2 - MAD
Description: To assess cumulative amount of analyte excreted from 0 to 24 hours (CumAe0-24) for Part 2
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
nmol | 2295 (638.1) [0.52 to 1.53] | 5540 (1305) [0.53 to 2.00] | 11390 (2415) [0.52 to 1.50] | 4002 (1402) | 11960 (4665) | 24970 (8075)

26. Secondary Outcome: Effect of Food on Absorption AZD7986 by Assessment of the Area Under the Plasma Concentration Versus Time Curve, From Time Zero to the Time of the Last Quantifiable Concentration (AUC(0-last)) for Part 1a and 1b - SAD
Description: To assess the effect of food by evaluating the area under the plasma concentration versus time curve, from time zero to the time of the last quantifiable analyte concentration (AUC(0-last)) for Part 1a (fasted state) and 1b (fed state) - SAD
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 hours); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h·nmol/L
Arm/Group | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 5
h·nmol/L | 12430 (18.3) | 10790 (20.2)

27. Secondary Outcome: Effect of Food on Absorption AZD7986 by Assessment of the Area Under Plasma Concentration-time Curve From Zero Extrapolated to Infinity (AUC) for Part 1a and 1b - SAD
Description: To assess the effect of food by evaluating the area under plasma concentration-time curve from zero extrapolated to infinity (AUC) for Part 1a (fasted state) and 1b (fed state) - SAD. AUC was estimated by AUC(0 last) + Clast/λz where Clast was the last observed quantifiable concentration.
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 hours); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h·nmol/L
Arm/Group | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 5
h·nmol/L | 13230 (19.6) | 11550 (22.6)

28. Secondary Outcome: Effect of Food on Absorption AZD7986 by Assessment of the Observed Maximum Plasma Concentration (Cmax) for Part 1a and 1b - SAD
Description: To assess the effect of food by evaluating the observed maximum plasma concentration (Cmax) for Part 1a (fasted state) and 1b (fed state) - SAD. Cmax was taken directly from the individual concentration-time curve
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 hours); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 5
nmol/L | 668.1 (26.7) | 434.8 (14.0)

29. Secondary Outcome: Effect of Food on Absorption AZD7986 by Assessment of the Time to Reach Maximum Observed Concentration (Tmax) for Part 1a and 1b - SAD
Description: To assess the effect of food by evaluating the time to reach maximum observed concentration (tmax) for Part 1a (fasted state) and 1b (fed state) - SAD; tmax was taken directly from the individual concentration-time curve
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 hours); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour
Arm/Group | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 5
Hour | 0.75 (26.7) [0.53 to 1.50] | 4.00 (14.0) [3.00 to 4.98]

30. Secondary Outcome: Effect of Food on Absorption AZD7986 by Assessment of the Apparent Terminal Elimination Half-life (t½.λz) for Part 1a and 1b - SAD
Description: To assess the effect of food by evaluating the half life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½.λz) for Part 1a (fasted state) and 1b (fed state) - SAD
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 hours); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 5
Hour | 23.80 (3.328) [0.53 to 1.50] | 24.24 (4.259) [3.00 to 4.98]

31. Secondary Outcome: Effect of Food on Absorption AZD7986 by Assessment of the Mean Residence Time (MRT) for Part 1a and 1b - SAD
Description: To assess the effect of food by evaluating the mean residence time (MRT) for Part 1a (fasted state) and 1b (fed state) - SAD
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 hours); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 5
Hour | 32.15 (5.003) [0.53 to 1.50] | 33.73 (6.429) [3.00 to 4.98]

32. Secondary Outcome: Effect of Food on Absorption AZD7986 by Assessment of the Apparent Clearance (CL/F) for Part 1a and 1b - SAD
Description: To assess the effect of food by evaluating the apparent clearance (CL/F) for Part 1a (fasted state) and 1b (fed state) - SAD; CL/F for parent drug was estimated as dose divided by AUC
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 hours); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litre/Hour
Arm/Group | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 5
Litre/Hour | 6.395 (1.281) [0.53 to 1.50] | 7.363 (1.810) [3.00 to 4.98]

33. Secondary Outcome: Effect of Food on Absorption AZD7986 by Assessment of the Apparent Volume of Distribution (Vz/F) for Part 1a and 1b - SAD
Description: To assess the effect of food by evaluating the apparent volume of distribution (Vz/F) for Part 1a (fasted state) and 1b (fed state) - SAD; Vz/F at terminal phase (extravascular administration) was estimated by dividing the apparent clearance (CL/F) by λz
Time Frame: At Day 1 (Pre-dose, 0.5, 1, 2, 3, 4, 5, 7, 8, 9, 12 hours); Day 2 (24 h); Day 3 (48 h); Day 4 (72 h) and Day 5 (96 h)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | AZD7986 35mg - Part 1a (Fasted State) - SAD | AZD7986 35mg - Part 1b (Fed State) - SAD
Number analyzed (Participants) | 6 | 5
Litre | 215.8 (29.62) | 249.5 (24.96)

34. Secondary Outcome: Assessment of Mean Normalized Relative Neutrophil Elastase (NE) Activity in All Cohorts of Part 2
Description: Absolute neutrophil count (ANC) was evaluated as part of the safety laboratory assessments and to evaluate the pharmacodynamics (PD) marker
Time Frame: At Day 16, 21 ((last dosing day in Cohort 1), 25, 28 (last sampling day in Cohort 1 and last dosing day in Cohorts 2 and 3), 32, 38, 41 and 52
Population: All participants who receiving at least 1 dose of AZD7986 or placebo and who had at least 1 pre-dose and 1 post-dose measurement for either NE (NE1 or NE2), and who had no major protocol deviations thought to impact on the analysis of the PD data
Measure: Mean (Standard Deviation); unit: Percentage change in NE activity
Groups:
- AZD7986 10mg - Part 2 - MAD: Participants received single dose of oral solution of AZD7986 10mg on Day 1 and daily dosing on Days 21 or 28 in fasted state.
- AZD7986 25mg - Part 2 - MAD: Participants received single dose of oral solution of AZD7986 25mg on Day 1 and daily dosing on Days 21 or 28 in fasted state.
- AZD7986 40mg - Part 2 - MAD: Participants received single dose of oral solution of AZD7986 40mg on Day 1 and daily dosing on Days 21 or 28 I fasted state.
Arm/Group | AZD7986 10mg - Part 2 - MAD | AZD7986 25mg - Part 2 - MAD | AZD7986 40mg - Part 2 - MAD | Placebo - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 12
Percentage change in NE activity
  Day 16 | -7.53 (11.59) | -28.25 (22.33) | -28.10 (16.87) | 7.39 (13.06)
  Day 21: number analyzed (Participants) | 5 | 7 | 10 | 10
  Day 21 | -26.13 (3.116) | -36.73 (11.76) | -52.31 (14.90) | 1.39 (20.14)
  Day 25: number analyzed (Participants) | 6 | 7 | 9 | 12
  Day 25 | -30.15 (8.412) | -40.06 (6.609) | -59.02 (11.77) | -5.15 (14.14)
  Day 28: number analyzed (Participants) | 6 | 7 | 7 | 8
  Day 28 | -39.22 (9.141) | -45.05 (8.304) | -55.24 (9.087) | -16.36 (22.03)
  Day 32: number analyzed (Participants) | 6 | 7 | 9 | 9
  Day 32 | NA (NA) — NA: not applicable. | -53.35 (8.292) | -46.29 (37.55) | -6.216 (14.28)
  Day 38: number analyzed (Participants) | 6 | 7 | 10 | 9
  Day 38 | NA (NA) — NA: not applicable. | -54.42 (6.800) | -65.44 (7.556) | -19.51 (10.74)
  Day 41: number analyzed (Participants) | 6 | 7 | 10 | 9
  Day 41 | NA (NA) — NA: not applicable. | -53.46 (9.774) | -62.56 (8.324) | -18.14 (15.62)
  Day 52: number analyzed (Participants) | 6 | 7 | 10 | 9
  Day 52 | NA (NA) — NA: not applicable. | -17.73 (18.07) | -21.31 (18.07) | -20.98 (15.32)

35. Secondary Outcome: Assessment of Absolute Neutrophil Count (ANC) in All Cohorts of Part 2
Description: as for outcome 34
Time Frame: At Day 12 (pre-dose, 6 hours and 12 hours)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: 10^9 neutrophils/L
Arm/Group | AZD7986 10mg - Part 2 - MAD | AZD7986 25mg - Part 2 - MAD | AZD7986 40mg - Part 2 - MAD | Placebo - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 12
10^9 neutrophils/L
  Day 12, Pre-dose: number analyzed (Participants) | 6 | 8 | 10 | 11
  Day 12, Pre-dose | 2.757 (0.4178) | 2.881 (0.5222) | 2.560 (0.9108) | 2.945 (0.7966)
  Day 12, 6 h: number analyzed (Participants) | 6 | 8 | 10 | 9
  Day 12, 6 h | NA (NA) — NA: not applicable. Not assessed for AZD7986 10 mg. | 3.401 (1.049) | 3.129 (0.7210) | 3.402 (1.178)
  Day 12, 12 h: number analyzed (Participants) | 6 | 8 | 10 | 9
  Day 12, 12 h | NA (NA) — NA: not applicable. Not assessed for AZD7986 10 mg. | 3.454 (0.7448) | 3.460 (0.5248) | 3.247 (0.7622)

36. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of Urine PK (Percentage of Dose Excreted Unchanged Into the Urine From 0 to 24 Hours (Cumfe0-24)) Parameter for Part 2 - MAD
Description: To assess percentage of dose excreted unchanged into the urine from 0 to 24 hours (Cumfe0 24) for Part 2
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of dose excreted unchanged
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
Percentage of dose excreted unchanged | 9.650 (2.683) [0.75 to 1.50] | 9.319 (2.195) [NA to NA] | 11.98 (2.539) [NA to NA] | 16.83 (5.894) | 20.12 (7.847) | 26.25 (8.489)

37. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of Urine PK (Renal Clearance From 0 to 24 Hours (CLR0-24)) Parameter for Part 2 - MAD
Description: To assess renal clearance from 0 to 24 hours (CLR0-24) for Part 2
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
Liter/hour | 1.784 (0.4606) [0.75 to 1.50] | 1.685 (0.3441) [NA to NA] | 1.782 (0.3841) [NA to NA] | NA (NA) — NA - Not applicable | NA (NA) — NA - Not applicable | NA (NA) — NA - Not applicable

38. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of Urine PK (Cumulative Amount of Analyte Excreted From 0 to 48 Hours (CumAe0-48)) Parameter for Part 2 - MAD
Description: To assess Cumulative amount of analyte excreted from 0 to 48 hours (CumAe0-48)) for Part 2
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
nmol | NA (NA) — NA - Not applicable. Not assessed for Day 1 | NA (NA) — NA - Not applicable. Not assessed for Day 1 | NA (NA) — NA - Not applicable. Not assessed for Day 1 | 6525 (2684) | 18680 (8765) | 36160 (12030)

39. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of Urine PK (Percentage of Dose Excreted Unchanged Into the Urine From 0 to 48 Hours (Cumfe0 48)) Parameter for Part 2 - MAD
Description: To assess Percentage of dose excreted unchanged into the urine from 0 to 48 hours (Cumfe0 48) for Part 2
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of dose excreted unchanged
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
Percentage of dose excreted unchanged | NA (NA) — NA - Not applicable. Not assessed for Day 1 | NA (NA) — NA - Not applicable. Not assessed for Day 1 | NA (NA) — NA - Not applicable. Not assessed for Day 1 | 27.44 (11.29) | 31.42 (14.74) | 38.01 (12.65)

40. Primary Outcome: Rate and Extent of Absorption of AZD7986 by Assessment of Urine PK (Renal Clearance From 0 to 48 Hours (CLR0-48)) Parameter for Part 2 - MAD
Description: To assess Percentage of dose excreted unchanged into the urine from 0 to 48 hours (Cumfe0 48) for Part 2
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | AZD7986 10mg - Day 1 - Part 2 - MAD | AZD7986 25mg - Day 1 - Part 2 - MAD | AZD7986 40mg - Day 1 - Part 2 - MAD | AZD7986 10mg - Day 21 - Part 2 - MAD | AZD7986 25mg - Day 28 - Part 2 - MAD | AZD7986 40mg - Day 28 - Part 2 - MAD
Number analyzed (Participants) | 6 | 8 | 10 | 6 | 7 | 10
Liter/hour | NA (NA) — NA - Not applicable. Not assessed for Day 1 | NA (NA) — NA - Not applicable. Not assessed for Day 1 | NA (NA) — NA - Not applicable. Not assessed for Day 1 | 1.508 (0.438) | 1.618 (0.5085) | 1.527 (0.3418)

ADVERSE EVENTS:
Time Frame: Part 1a and 1b: Day -1, Day 1 to Day 3 (spontaneous, at pre-dose, 3, 12, 24, 48 and 72 hours [h] post-dose), Day 4, Day 5 and follow-up (7-10 days after dosing [not for participants included in Part 1b]); Part 2: Day -1, Day 1 to Day 21/28 and follow-up
Description: All randomized participants who received at least 1 dose of IMP were included in the safety analysis.
  Adverse events (AEs - serious / non-serious), an undesirable medical condition occurring at any time after the participant had signed informed consent, including run-in or washout periods, even if no specific treatment has been administered.
Arm/Group | Part 1a (Fasted State) - Single Ascending Dose (SAD) | Part 1b (Fed State) - SAD | Part 2 - Multiple Ascending Dose (MAD) | Placebo - Part 1a (Fasted State)- SAD | Placebo - Part 1b (Fed State) - SAD | Placebo - Part 2 - MAD
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/5 | 0/24 | 0/15 | 0/3 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/5 | 0/24 | 0/15 | 0/3 | 0/12
Other Adverse Events (participants affected / at risk) | 8/30 | 2/5 | 23/24 | 8/15 | 1/3 | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1a (Fasted State) - Single Ascending Dose (SAD) (N=30) | Part 1b (Fed State) - SAD (N=5) | Part 2 - Multiple Ascending Dose (MAD) (N=24) | Placebo - Part 1a (Fasted State)- SAD (N=15) | Placebo - Part 1b (Fed State) - SAD (N=3) | Placebo - Part 2 - MAD (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 6 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 1 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 2 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 3 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Systolic hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (General disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.